CLINICAL TRIAL: NCT05576077
Title: A Phase 1b Study of TBio-4101 (Autologous Selected and Expanded Tumor-Infiltrating Lymphocytes [TIL]) and Pembrolizumab in Patients With Advanced Solid Tumor Malignancies (STARLING)
Brief Title: A Study of TBio-4101 (TIL) and Pembrolizumab in Patients With Advanced Solid Tumors
Acronym: STARLING
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Turnstone Biologics, Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBio-4101-001
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Colorectal Cancer; Uveal Melanoma; Cutaneous Melanoma; Non-Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: MSS-CRC; TIL; Tumor infiltrating lymphocyte; TNBC; HR+ Breast; ER+ Breast; MSI-CRC; personalized medicine; ocular melanoma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Uveal Melanoma; Melanoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — Toll-Like Receptor 1; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Patients enrolled into a Cohort based on malignancy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Breast Cancer (Experimental): Patients with locally advanced or metastatic breast cancer that has failed or is intolerant to standard of care therapies. Includes, HER2+, HER 2-, TNBC.
  Interventions: Biological: TBio-4101; Drug: Pembrolizumab
- Colorectal carcinoma (Experimental): Patients with advanced, metastatic colorectal adenocarcinoma who have failed or are intolerant to at least one line of therapy that included either irinotecan or oxaliplatin.
  Interventions: Biological: TBio-4101; Drug: Pembrolizumab
- Uveal Melanoma (Experimental): Patients with advanced, metastatic uveal melanoma.
  Interventions: Biological: TBio-4101; Drug: Pembrolizumab
- Cutaneous Melanoma (Experimental): Patients with cutaneous melanoma who have experienced disease progression following a PD-1 or PD-L1 inhibitor.
  Interventions: Biological: TBio-4101; Drug: Pembrolizumab
- Non-Small Cell Lung Cancer (Experimental): Patients with non-small cell lung cancer who have experienced disease progression following platinum containing chemotherapy and/or PD-1 or PD-L1 inhibitor.
  Interventions: Biological: TBio-4101; Drug: Pembrolizumab
- Head and Neck Squamous Cell Carcinoma (Experimental): * Patients with head and neck squamous cell carcinoma who have received no prior therapy for metastatic disease
  * Patients with head and neck squamous cell carcinoma who are PD-1/PD-L1 inhibitor naïve at the time of TIL harvest and will be treated with TBio-4101 at the time of progression, inadequate response or intolerance to the PD-1/PD-L1 inhibitor-based standard of care regimen given on study.
  Interventions: Biological: TBio-4101; Drug: Pembrolizumab

INTERVENTIONS:
Biological: TBio-4101 — TBio-4101 is an autologous selected and expanded tumor infiltrating lymphocyte (TIL) product generated following ex vivo expansion of tumor reactive TIL population found in tumor harvest. After preparation with non-myeloablative lymphodepletion chemotherapy (cyclophosphamide and fludarabine) followed by low dose radiation,TBio-4101, and IL-2.
  Other Names: TIL, autologous, tumor-reactive, T-cell product
Drug: Pembrolizumab — Pembrolizumab will be administered after TIL infusion and continue every 3-6 weeks for up to 2 years.
  Other Names: Keytruda

SUMMARY:
A multicenter trial to investigate TBio-4101, an autologous, neoantigen-selected, tumor-reactive TIL product, in patients with advanced solid malignancies.

DETAILED DESCRIPTION:
This is a Phase 1 study to investigate TBio-4101. TBio-4101 is an autologous tumor infiltrating lymphocyte (TIL) therapy that utilizes tumor specific antigens to select, sort, and expand patient-specific tumor-reactive T-cells to be reinfused into the patient. The adoptive cell therapy is further enhanced through the use of non-myeloablative chemotherapy prior to TIL infusion, followed by the TIL plus IL-2 infusion. Low-dose radiation therapy is administered prior to and after TIL plus IL-2 infusion. Pembrolizumab is provided after the resolution of IL-2 toxicities. The trial is open to solid tumors of varying tumor mutational burdens.

ELIGIBILITY:
Key Inclusion Criteria:

* Advanced or metastatic breast carcinoma, colorectal adenocarcinoma, uveal melanoma, cutaneous melanoma, non-small cell lung cancer, or head and neck squamous cell carcinoma that has failed or is refractory to standard of care therapy
* Have at least one target lesion that can be used for response assessments and have at least 1 tumor amenable for tissue harvest for TIL manufacturing.
* ECOG performance status of 0 or 1
* Demonstrate adequate organ function
* Additional inclusion criteria exist

Key Exclusion Criteria:

* Known additional malignancy that is progressing or has required active treatment within the past 3 years
* Diagnosis of immunodeficiency or receiving chronic systemic steroid therapy or any other form of immunosuppressive
* Currently infected with HIV Type 1 and Type 2, hepatitis B virus (HBV), hepatitis C virus (HCV), treponema pallidum (e.g., syphilis), West Nile virus (WNV), Human T-lymphotropic virus types 1 or II (HTLV I/II), or cytomegalovirus (CMV)
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable
* Serious cardiac condition, such as uncontrolled hypertension, concurrent congestive heart failure, prior history of Class III/IV cardiac disease (New York Heart Association [NYHA]), history of cardiac ischemia within the past 6 months, or prior history of cardiac arrhythmia requiring treatment. Patients who are > 60 years of age must undergo cardiology clearance exam and cardiac stress test.
* Prior cell therapy or organ transplant
* History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, IL-2, or pembrolizumab, or any of their constituents
* LVEF ≤ 45%
* FEV1 ≤ 60% of predicted value and DLCO (corrected) < 60% of predicted value
* Chronic anti-coagulant therapy that cannot either be discontinued or temporarily changed
* Additional exclusion criteria exist

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 25 months
  The incidence of treatment-emergent adverse events will be tabulated using NCI CTCAE v5.0

SECONDARY OUTCOMES:
Proportion of patients with a response (ORR) | 25 months
  Percentage of all patients and within each cancer indication with a CR or PR as assessed by the independent central radiologist using RECIST 1.1 and iRECIST
Estimated Disease Control Rate (DCR) | 25 months
  Portion of patient whose best response is a CR, PR, or stable disease (SD) as assessed by the independent central radiologist using RECIST v1.1 and iRECIST
Estimated Duration of Response (DoR) | 25 months
  Duration of response, as measured in weeks, that patients with a CR or PR have no progressed (PD), as assessed by the independent central radiologist using RECIST v1.1 and iRECIST,

CONTACTS AND LOCATIONS:
Overall Officials: Ines Verdon, MD, Study Director — Turnstone Biologics, Corp.
Locations (13):
- United States (11):
  - University of California Irvine, Irvine, California
  - Memorial Healthcare System, Hollywood, Florida
  - University of Miami, Miami, Florida
  - Orlando Health, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Providence Cancer Institute, Portland, Oregon
  - Allegheny Research Institute, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Montreal University Hospital Center, Montreal, Quebec